CLINICAL TRIAL: NCT01331642
Title: Biomarker for Gaucher Disease an International, Multicenter, Epidemiological Protocol
Brief Title: Biomarker for Gaucher Disease: BioGaucher (BioGaucher)
Acronym: BioGaucher
Status: Withdrawn | Type: Observational
Why Stopped: Transition to BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BG 06-2018
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Splenomegaly; Hepatomegaly
Keywords: Gaucher Disease; Biomarker
MeSH Terms: conditions — Splenomegaly; Hepatomegaly; Gaucher Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of Mass-spectrometry, maximal 10 ml blood will be taken via using a dry blood spot filter card and will be ana-lysed. (Optionally, also 10 ml urine will be taken via urine-collection tube). To proof the correct Gaucher diagnosis in those patients where up to the enrollment in the study no genetic testing has been done, sequencing of Gaucher will be done.
  The analyses will done at:
  Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Patients with Gaucher disease or high-grade suspicion for Gaucher disease

SUMMARY:
Development of a new mass spectrometry-based biomarker for the early and sensitive diagnosis of Gaucher Disease from blood (plasma)

DETAILED DESCRIPTION:
Gaucher disease (GD) is an autosomal recessive hereditary lysosomal storage disorder. Occurrence of the disease is due to a hereditary deficiency of the Glucocerebrosidase, a lysosomal enzyme which divides Glucocerebroside into Glucose and Ceramides. The unmetabolised Glucocerebrosides are stored throughout the whole reticulo-endothelial system. Accumulation of Glycolipid-enriched macrophages establishes a pathoanatomical phenomenon, the so-called Gaucher cells, which can be verified by light microscopy of affected tissues. Activation markers of the macrophages, like the enzyme Chitotriosidase or CCL18, are parameters which follow the course of GD.

Gaucher disease is the most frequently inherited Sphingolipidosis in the general population, and in Ashkenazi Jews, in who the prevalence is much higher (1:450). The gene which codes the Glucocerebrosidase is on the long arm of chromosome 1 and covers 11 exons. So far, more than 200 different mutations in Gaucher patients have been described, mostly missense mutations. In addition, frame-shift- and splice-site-mutations have been detected, as well as insertions and deletions. More frequent mutations are N370S, L444P, IVS2+1G>A, c.84insG, R463C and R496H.

The clinical appearance is heterogeneous. The classical phenotype is characterised by visceral organ (Hepatosplenomegaly) and skeleton system (Bone marrow infiltrates up to bone infarcts and pathological fractures) affection. Moreover, consecutive blood cell count changes, Anemia and Thrombocytopenia are reported.

A serious distinction lies in the appearance of neurological manifestations (myoclonus epilepsy, hydrocephalus, ocular movement disturbances). There is discussion on whether the classification into the typical three disease types (type1: non-neuronopathic progress form, type2: acute neuronopathic progress form, type3: chronic neuronopathic progress form) is still up-to-date, since it does not sufficiently reflect the reality of the clinical presentation. A clear genotype-phenotype relationship does not exist. The same DNA mutations are detected in patients with pronounced differences in disease progression. The exception is the mutation N370S, which has so far been detected in connection with only visceral progress forms (type1). At least the outcome of the non-neuronopathic disorder cases could be improved by the introduction and general availability of enzyme therapy. Under this kind of therapy there is a reduction of liver and spleen size as well as a normalization of the haemogram parameters.

New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood (plasma) of affected patients that allow to diagnose in the future the disease earlier, with a higher sensitivity and specificity. In a pilot study lyso-glycosylsphingosine has been determined as a sensitive and specific biomarker (see attached manuscript). This is a metabolic product likely to be involved in the pathophysiology of the disease. Therefore it is the goal of the study to validate this new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and there-by with an earlier treatment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained from the patient or the parents before any study related procedures.
* Patients of both gender from the first day of life
* The patient has a diagnosis of Gaucher disease or high-grade suspicion for Gaucher disease
* High-grade suspicion present, if one or more criteria are valid:

  1. - Positive family anamnesis for Gaucher disease
  2. - Splenomegaly without identifiable cause
  3. - Hepatomegaly without identifiable cause
  4. - Anemia or thrombocytopenia without identifiable cause
  5. - CNS involvement without identifiable cause

Exclusion Criteria:

* No Informed consent from the patient or the parents before any study related pro-cedures
* No diagnosis of Gaucher disease or no valid criteria for high-grade suspicion of Gaucher disease

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Gaucher disease or high-grade suspicion for Gaucher disease
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Sequencing of the Gaucher disease related gene | 4 weeks
  Next-Generation Sequencing (NGS) of the GBA gene will be performed. The mutation will be confirmed by Sanger sequencing.

SECONDARY OUTCOMES:
The Gaucher disease specific biomarker candidates finding | 24 months
  The quantitative determination of small molecules (molecular weight 150-700 kD, given as ng/μl) within a dried blood spot sample will be validated via liquid chromatography multiple reaction-monitoring mass spectrometry (LC/MRM-MS) and compared with a merged control cohort. The statistically best validated molecule will be considered as a disease specific biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (4):
- Centogene AG, Rostock, Germany
- India (2):
  - Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala
  - Navi Mumbai Institute of Research In Mental And Neurological Handicap (NIRMAN), Mumbai
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided